CLINICAL TRIAL: NCT00574652
Title: ANRS HC 21 VASCU IL-2, Evaluation of the Cellular Immune Response, Clinical Efficacy and Tolerance After IL-2 Therapy in HCV-related Vasculitis Patients, Resistant to Conventional Therapy.
Brief Title: Evaluation of Clinical Efficacy and Immunologic Response After IL-2 Therapy in HCV-related Vasculitis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-004039-31; ANRS HC 21 Vascu-IL2
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Cryoglobulinemia Vasculitis
Keywords: HCV+; cryoglobulinemia; Vasculitis; IL-2 treatment; safety and efficacy
MeSH Terms: conditions — Cryoglobulinemia; Vasculitis | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): it is a single arm study
  Interventions: Drug: Proleukin

INTERVENTIONS:
Drug: Proleukin — 3 millions IU/day from day 1 to 5 every 21 days will be carried out at W1, W3, W6, and W9)
  Other Names: Aldesleukin; Novartis Pharma S.A.S

SUMMARY:
A systemic Vasculitis is found in 5 to 10% of HCV infected patients with mixed cryoglobulinemia (MC). It mainly involves the skin, peripheral nerve and the kidney and may be life threatening. Twenty to 30% of HCV-MC Vasculitis patients are resistant to conventional therapy (i.e. antiviral therapy and/or immunosuppressors) and still have an active disease. Thus, new therapeutic approaches are necessary in such patients. We recently described a regulatory T cell (Treg) deficiency in HCV-related Vasculitis patients. Immunomodulatory effects of interleukin-2 (IL-2) are well established, notably the preferential expansion of Treg able to suppress inflammatory responses mediated by CD4+ and CD8+ T cells.

DETAILED DESCRIPTION:
A systemic Vasculitis is found in 5 to 10% of HCV infected patients with mixed cryoglobulinemia (MC). It mainly involves the skin, peripheral nerve and the kidney and may be life threatening (15% of death). Twenty to 30% of HCV-MC Vasculitis patients are resistant to conventional therapy (i.e. antiviral therapy and/or immunosuppressors) and still have an active disease. An antiviral therapy with Peg-interféron is generally prescribed to control Vasculitis lesions and to slow down the hepatic fibrosis progression. Thus, new therapeutic approaches are necessary in such patients. We recently described a CD4+ CD25+ regulatory T cell (Treg) deficiency in HCV-related Vasculitis patients. Immunomodulatory effects of interleukin-2 (IL-2) are well established, notably the preferential expansion of Treg able to suppress inflammatory responses mediated by CD4+ and CD8+ T cells.

Objective : To evaluate the cellular immune response after IL-2 therapy in HCV-MC Vasculitis patients, resistant to conventional therapy.

Methods : This is an open prospective phase I/II trial. Four cycle of subcutaneous IL-2 therapy (3 millions IU/day from day 1 to 5 every 21 days will be carried out at W1, W3, W6, and W9). The first cure will be carried out with half-dose of IL-2 (1.5 millions IU/day) in the hospital. If the tolerance is satisfactory, the later cures will be done ambulatory. All patients will be followed after IL-2 therapy (S11 to S37).

End points :

1. Clinical tolerance: Absence of Vasculitis flare during and after IL-2 therapy.
2. Immunologic follow-up of Treg and of HCV cellular immune response before, during and after IL-2 therapy.
3. Clinical efficacy: follow-up of clinical manifestations of HCV-MC Vasculitis during and after IL-2 therapy.

Schedule : Duration of patients' inclusion period is estimated 18 months. Duration of therapy and follow-up is estimated 9 months. Analysis of data will last 7 months. Overall duration: 34 months

ELIGIBILITY:
Inclusion Criteria:

1. HCV+ patients with cryoglobulinemia Vasculitis
2. resistant to conventional therapy (i.e. antiviral therapy and/or immunosuppressors).
3. Vasculitis is defined according to international criteria: chronic HCV infection (HCV RNA+),
4. serum cryoglobulin superior or equal to 0.05g/l in at least two determinations,
5. presence of the triad purpura-arthralgia-asthenia and/or biopsy proven Vasculitis (kidney, nerve or skin).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Immunologic follow-up of Treg and of HCV cellular immune response before, during and after IL-2 therapy | 9 months

SECONDARY OUTCOMES:
Clinical tolerance: Absence of Vasculitis flare during and after IL-2 therapy | 9 months
Clinical efficacy: follow-up of clinical manifestations of HCV-MC | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Cacoub, MD, PHD, Principal Investigator — Hôpital de la Pitié, 83 Bd de l'Hôpital 75651 Paris cedex 13
Locations (1):
- Hôpital de la Pitié, Paris, France

REFERENCES:
- [Derived] Saadoun D, Rosenzwajg M, Joly F, Six A, Carrat F, Thibault V, Sene D, Cacoub P, Klatzmann D. Regulatory T-cell responses to low-dose interleukin-2 in HCV-induced vasculitis. N Engl J Med. 2011 Dec 1;365(22):2067-77. doi: 10.1056/NEJMoa1105143. PMID 22129253